CLINICAL TRIAL: NCT03409497
Title: Effects of Grape Juice With Breakfast on Glycemia and Cognitive Function in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Welch's Food Corporation (Unknown)
Responsible Party: Principal Investigator, Richard Mattes, Principle Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 055-049
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2019-08

CONDITIONS: Glycemic Response; Appetitive Behavior
MeSH Terms: conditions — Appetitive Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Concord Grape Juice (Active Comparator): Concord Grape Juice
  Interventions: Other: Concord Grape Juice
- Low flavonoid low essence beverage (Sham Comparator): Low flavonoid low essence beverage
  Interventions: Other: Low flavonoid low essence beverage
- Low flavonoid beverage (Sham Comparator): Low flavonoid beverage
  Interventions: Other: Low flavonoid beverage

INTERVENTIONS:
Other: Concord Grape Juice — Concord Grape Juice
  Arms: Concord Grape Juice
Other: Low flavonoid low essence beverage — Low flavonoid low essence beverage
  Arms: Low flavonoid low essence beverage
Other: Low flavonoid beverage — Low flavonoid beverage
  Arms: Low flavonoid beverage

SUMMARY:
Assess the impact of 100% grape juice with a meal on postprandial glycemic response and subsequent appetite, food intake and cognitive function.

DETAILED DESCRIPTION:
Investigators earlier studies and published literature suggest that the phenolic content and strong flavor intensity of 100% Concord grape juice hold potential beneficial effects on blood sugar levels. Investigators aim to better understand the consumption of 100% grape juice with a meal modifies appetite and glycemia acutely and over the day using a 24 hour glucose monitor.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25.0-34.9 kg/m2
* Willingness to eat all test foods
* Low consumer of tea and coffee, willingness to refrain from both during the 48 hours prior to test days and on the test day
* Fasting blood glucose below 6.1mmol/l via capillary finger-stick blood sample using a SureStep glucometer (Lifescan, Milpitas, CA)

Exclusion Criteria:

* Taking medications known to affect glycemia, lipid metabolism or appetite
* Body weight fluctuation of >5kg in the past 3 months
* Taking vitamin or other supplements
* Smokers
* Acute or Chronic disease

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
change in blood glucose over 24 hours | 24 hours
  samples taken every 5 minutes for 24 hours by a continuous glucose monitor

SECONDARY OUTCOMES:
Appetite | 24 hours
  Questionnaire on hunger, fullness, desire to eat, prospective consumption, thirst taken hourly on same day as grape juice intervention

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Coelho OGL, Alfenas RCG, Debelo H, Wightman JD, Ferruzzi MG, Mattes RD. Effects of Concord grape juice flavor intensity and phenolic compound content on glycemia, appetite and cognitive function in adults with excess body weight: a randomized double-blind crossover trial. Food Funct. 2021 Nov 15;12(22):11469-11481. doi: 10.1039/d1fo02049h. PMID 34698750